CLINICAL TRIAL: NCT07079293
Title: Extended Platelet- Rich Fibrin Membrane Combined With Vestibular Incision Subperiosteal Tunnel Access Technique as a New Treatment Modality for Localized Gingival Recession (Clinical Comparative Study)
Brief Title: Extended Platelet- Rich Fibrin Membrane Combined With Vestibular Incision Subperiosteal Tunnel Access Technique to Treat Localized Gingival Recession
Acronym: alb prf REC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0801024OM
Record Dates: First submitted 2025-07-13; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Gingival Recession, Localized
Keywords: CTG; alb prf; extended prf; e prf; G.REC; VISTA; RT1; CAIRO
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (control group): Connective Tissue Graft to treat patient had RT1 Gingival Recession (Experimental): 15 patients will be treated with free gingival graft harvested from the hard palate then de-epithelized outside the oral cavity to be used in conjunction with VISTA technique for treatment of type 1 recession (RT1).
  Interventions: Procedure: Harvesting of Free Gingival Graft and preparation of CTG; Procedure: VISTA technique
- Group 2 (study group): Alb prf membrane to treat patient had RT1 Gingival Recession (Experimental): 15 patients will be treated with extended platelet-rich fibrin (e-PRF) (Alb prf) membrane to be used in conjunction with VISTA technique for treatment of type 1 recession (RT1).
  Interventions: Other: Preparation of Extended PRF; Procedure: VISTA technique

INTERVENTIONS:
Other: Preparation of Extended PRF — Whole blood (10 mL) will be centrifuged at 700 g for 8 minutes. The upper layer (yellow layer) shows the liquid plasma layer. The most upper layer of platelet- poor plasma (PPP) will be collected in a syringe. then PPP will be heated in a heat block device at 75°C for 10 minutes and thereafter cooled to room temperature for approximately 2 minutes. An injectable albumin gel will then be prepared. Then the liquid platelet-rich layer (liquid-PRF) including the buffy coat layer with accumulated platelets and leukocytes, will be collected in a separate syringe. The albumin gel and native liquid PRF will then be thoroughly mixed by utilizing a female-female luer lock connector. Now injectable e-PRF in final form is ready to be used .
  Arms: Group 2 (study group): Alb prf membrane to treat patient had RT1 Gingival Recession
Procedure: Harvesting of Free Gingival Graft and preparation of CTG — The region distal from the canines, commencing at least 2 mm from the gingival margin with a width of 5-8 mm and a desirable length to cover the entire recipient site is an ideal site for harvesting a FGG from the hard palate for root coverage. Harvesting of FGG is performed as follows: The graft is prepared by outlining with two parallel longitudinal incisions that are interconnected with vertical incisions. Graft deliberation is initiated along the paramarginal incision in a split-thickness fashion with a goal of removing an FGG of 1.5-2-mm thickness without touching the periosteum. The harvested free gingival graft will be de-epithelialized to obtain an DFGG. The donor site wound will be covered by gel foam which will be sutured in place and then healing will occur by secondary intention .
  Arms: Group I (control group): Connective Tissue Graft to treat patient had RT1 Gingival Recession
Procedure: VISTA technique — Following Zadeh's (2011) protocol, under local anesthesia, a vestibular access incision is made depending on the treatment site (midline frenum for maxillary anterior, frenal area between canine and lateral incisor for maxillary posterior, and similar for mandibular regions). The incision passes through the periosteum to create a subperiosteal tunnel exposing the facial bone and root dehiscence. In the test group, the extended platelet-rich fibrin (e-PRF) membrane is inserted into the tunnel and secured to the flap with horizontal sutures; in the control group, a de-epithelialized free gingival graft (DFGG) is used similarly. Each tooth's facial enamel is briefly acid-etched, washed, and dried to attach vicryl sutures fixed with flowable composite resin to prevent apical relapse during healing. Finally, the access incision is closed and sutured with vicryl sutures

SUMMARY:
This study will be performed to clinically evaluate and compare the effectiveness of extended platelet-rich fibrin (e-PRF) membrane versus de-epithelized free gingival graft (DFGG) in combination with vestibular incision subperiosteal tunnel access (VISTA) in the treatment of localized Cairo gingival recession type 1 (RT1) defects.

The primary outcome of the present study will be the percentage of root coverage assessed after 6 months of surgical therapy whereas the secondary outcomes include the differences of gingival thickness, keratinized tissue width and dental hypersensitivity after 3 and 6 months.

DETAILED DESCRIPTION:
Gingival recession (GR) has been defined as the apical shift of the gingival margin in respect to the cementoenamel junction with concomitant exposure of the root surface in the oral cavity. Several etiological factors such as tissue phenotype, gingival thickness, brushing technique, non-carious and carious cervical lesions, and periodontal predisposition were identified for this condition, which may account for its relatively high incidence in the population .

When GR affects the esthetic area and is associated with dentinal hypersensitivity, exhibits a lack of an adequate band of keratinized tissue, or is concomitant with a carious or non-carious cervical lesion, treatment is often indicated. Indeed, the efficacy of surgical treatment for correction of GR defects has been extensively demonstrated with long-term stable outcomes .

With a broad variety of gingival recession cases with different clinical presentations, it is not always possible to classify all gingival recession defects according to one classification system. Several classifications have been proposed in literature to facilitate the diagnosis of gingival recessions. One of the most commonly used Cairo et al. classification (2011) which classified gingival recession based on the assessment of CAL at both buccal and interproximal sites into recession type 1, 2 and 3. This classification provides a simplified method of categorizing gingival recession and also emphasizes the role of interproximal attachment level, one of the important site-related prognostic factors .

Recession type 1 is characterized by gingival recession with no loss of interproximal attachment. Interproximal CEJ is clinically not detectable at both mesial and distal aspects of the tooth .

Several surgical techniques, such as guided tissue regeneration (GTR), subepithelial connective tissue graft procedure (SCTG), coronally advanced flap (CAF), laterally positioned flap, double papilla technique, semilunar pedicle flap, oblique rotated flap, tunnel technique (TUN), and surgical techniques based on modifications of these protocols have been proposed for the treatment of GR defects .

The subepithelial connective tissue graft (CTG) has been advanced as the "gold standard" for recession coverage around teeth . However, the limited amount of donor tissues, technique sensitivity and post-operative patient's discomfort are all considered as disadvantages for this technique .

Nowadays, patients' esthetic expectations and perception of the use of least traumatic surgeries have led to the development of minimally invasive techniques which not only obtain root coverage but also have a color match and tissue blending with adjacent tissues of the defect site .

The introduction of non-invasive techniques such as envelope and tunnel technique (TUN) had reduced the struggles in other invasive operations and provided good vascularity due to absence of the vertical releasing incision. Homa Zadeh in 2011 introduced a conservative modification in tunnel technique; vestibular incision subperiosteal tunnel access (VISTA) which preserves the papillary integrity and enhances patients' compliance .

Platelet concentration-based therapies were first used as fibrin adhesives in wound healing. Platelet-rich plasma, an autologous platelet concentration, was developed in 1998 as an enhancement factor for periodontal wound healing. Platelet-rich fibrin (PRF) is a second-generation autologous platelet concentration obtained without using any chemical substances such as anticoagulants and thrombin .

The effectiveness of autologous platelet concentration lies on the continuous release of multiple cytokines, such as transforming growth factor-β1 (TGF-β1), vascular endothelial growth factor (VEGF), insulin growth factor (IGF), platelet- derived growth factor-AB (PDGF-AB), and interleukin-1β (IL-1β) . Since the PRF preparation protocol does not require any anti-coagulants, wound healing cascade is not inhibited by anticoagulants and clot formation occurs naturally .

PRF has several advantages including high concentration of leukocytes which not only act in immune and antibacterial responses but also promote the wound-healing process. The PRF spontaneously forms a dense fibrin network that enables slower degradation rate and therefore delayed release of growth factors to the surrounding tissue during wound healing .

Platelet-rich fibrin (PRF) has been proposed as an autologous membrane with the advantages of host accumulation of platelets and leukocytes with entrapment of growth factors. However, limitations include its faster resorption properties (approximately 2 weeks). Interestingly, recent studies have demonstrated that by heating a liquid platelet-poor plasma (PPP) layer, the resorption properties of heated albumin (albumin gel) can be extended from 2 weeks to greater than 4 months (e- PRF) .

Given the encouraging effects of e-PRF in healing and regeneration of soft tissue with long-term release of growth factors, it is hypothesized that e-PRF might improve the outcomes obtained with vestibular incision subperiosteal tunnel access (VISTA) technique. To the best of the authors' knowledge, there is no controlled clinical study using VISTA combined with e-PRF for root coverage in localized Cairo type 1 recession defects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Cairo recession type 1 (RT1): Gingival recession with no loss of interproximal attachment. Interproximal CEJ is clinically not detectable at both mesial and distal aspects of the tooth (15).
2. No systemic diseases.
3. Non-smokers.
4. Good oral hygiene and no bleeding on probing.
5. No history of previous mucogingival surgeries.

Exclusion Criteria:

* 1. Detected interproximal alveolar bone loss.

  2. Pregnancy and lactating females

  3. Heavy smokers.

  4. Immunocompromised patients.

  5. Fixed prosthesis in the site that will be treated.

  6. Teeth with cervical caries, non-carious lesions or cervical fillings.

  7. Bad oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Root coverage percentage (RC%) | 6 months
  Root coverage percentage (%)

SECONDARY OUTCOMES:
Gingival thickness (GT) | 6 months
  measured using an endodontic spreader with stopper (#30) 2 mm apical to the buccal gingival margin under local anesthesia
Width of keratinized gingiva (WKG): | 6 months
  (measured at the mid buccal point from the free gingival margin to the mucogingival junction).
Sensitivity visual analogue scale (Sens VAS) | 6 months
  Dental hypersensitivity tested using the air spray and quantified by patients on a visual analogue scale (VAS) from 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University., Al Mansurah, Egypt